CLINICAL TRIAL: NCT01301560
Title: Randomized Phase III Trial of Stereotactic Radiosurgery (SRS) Versus Observation for Patients With Asymptomatic Cerebral Oligo-metastases in Non-small Cell Lung Cancer (NSCLC)
Brief Title: Chemotherapy With or Without Radiosurgery for Asymptomatic Oligo Brain Metastasis
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Samsung Medical Center (Other)
Responsible Party: Myung-Ju Ahn / Professor, Samsung Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2008-05-024
Record Dates: First submitted 2011-02-21; First posted 2011-02-23 (Estimated); Last update posted 2011-02-23 (Estimated); Status verified 2011-02

CONDITIONS: Nonsmall Cell Lung Cancer
Keywords: Asymptomatic brain metastasis; NSCLC; GKS
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Radiosurgery; Observation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Radiosurgery arm (Experimental): Radiosurgery before palliative chemotherapy
  Interventions: Radiation: Radiosurgery
- Observation arm (No Intervention): No radiotherapy or local treatment until specific symptoms or sign developed
  Interventions: Radiation: Observation

INTERVENTIONS:
Radiation: Radiosurgery — Gamma knife surgery for asymptomatic oligo-metastasis to brain from NSCLC
  Arms: Radiosurgery arm
Radiation: Observation — No local treatment
  Arms: Observation arm

SUMMARY:
The need of radiosurgery is controversial for asymptomatic oligo brain metastasis for non small cell lung cancer (NSCLC).

Therefore, the investigators do a randomized study comparing overall survival between two groups with or without radiosurgery for asymptomatic oligo brain metastasis before palliative chemotherapy for NSCLC.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed non-small cell lung cancer with synchronous brain metastases
2. One to 4 intraparenchymal brain metastases by contrast-enhanced MRI, meeting the following criteria:

   * Well circumscribed tumor(s) with brain edema Grade 0-1
   * Maximum diameter ≤ 3.0 cm
3. No prior surgical treatment or RT for brain metastases
4. No leptomeningeal metastases by MRI or cerebrospinal fluid evaluation
5. Patients without any symptoms or signs from brain metastases (RTOG neurologic functions status of 0)
6. Age, 18 and over
7. ECOG performance status 0-1
8. Written informed consent

Exclusion Criteria:

1. severe co-morbid illness and/or active infections
2. pregnant or lactating women
3. RTOG neurologic function status of 1~4
4. Uncontrollable extracranial metastases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 176 (Estimated)
Dates: Start 2008-06; Primary Completion 2013-05 (Estimated)

PRIMARY OUTCOMES:
overall survival | 1 year after the enrollment of the last patient

SECONDARY OUTCOMES:
Time to CNS progression | 1 year after the enrollment of the last patient

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung Medical Center, Seoul, South Korea

REFERENCES:
- [Derived] Lim SH, Lee JY, Lee MY, Kim HS, Lee J, Sun JM, Ahn JS, Um SW, Kim H, Kim BS, Kim ST, Na DL, Sun JY, Jung SH, Park K, Kwon OJ, Lee JI, Ahn MJ. A randomized phase III trial of stereotactic radiosurgery (SRS) versus observation for patients with asymptomatic cerebral oligo-metastases in non-small-cell lung cancer. Ann Oncol. 2015 Apr;26(4):762-768. doi: 10.1093/annonc/mdu584. Epub 2014 Dec 23. PMID 25538174